CLINICAL TRIAL: NCT00256217
Title: Phase II Chemoprevention Trial - Anastrozole in the DCIS and Early Invasive Breast Cancer in Postmenopausal Women
Brief Title: Chemoprevention Trial - Anastrozole in Ductal Carcinoma In Situ (DCIS) in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rita Sanghvi, Mehta (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Rita Sanghvi, Mehta, Dr. Rita Mehta, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 03-16 [HS# 2004-3681]; 2004-3681 (Other: University of California Irvine); NCI-2010-00361 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anastrozole (Experimental)
  Interventions: Drug: Anastrozole

INTERVENTIONS:
Drug: Anastrozole — 1 mg. oral every day for 2 - 4 weeks
  Other Names: ARIMIDEX

SUMMARY:
Breast cancer is one of the most common cancers seriously afflicting women in the United States. Of the one million incident cases that are reported annually there are approximately 193,000 new cases of breast cancer (Greenlee, 2001). Although significant advances have been made both in early detection and treatment of breast cancer, the impact of these on reduction in mortality has been modest (Peta, 2000). Furthermore, despite data implicating diet and other environmental risk factors, no lifestyle changes have yet been shown to significantly reduce the risk of breast cancer. Therefore, chemoprevention of breast cancer is a worthwhile approach to reduce the incidence of breast cancer.

There is every reason to believe that a detailed understanding of the initiation, promotion and growth of breast cancer will ultimately provide a rational strategy upon which to base prevention strategies. While the pathways of breast cancer development are not yet fully understood, a role for estrogens in breast cancer etiology has been well established.

While many pathways are involved in breast cancer etiology, including loss of tumor suppressor function by p53 or BRCA1 and gain of HER2 oncogene expression, their exact role in an individual patient's cancer development may vary.

Therefore, it may be advantageous to focus on a chemoprevention strategy that may have a more uniform impact on breast cancer development, such as estrogen exposure. Estrogen and its metabolites, both in the circulation and locally synthesized in the breast, are important in the pathogenesis of breast cancer. High levels of circulating estrogen in postmenopausal women have been associated with an increased risk of breast cancer (Clemons, 2001). Furthermore, local estrogen synthesis, i.e. aromatase activity, in the breast may also be important in the development of breast cancer.

DETAILED DESCRIPTION:
Specific Aim 1: We hypothesize that a proliferative marker Ki-67 is reduced in patients with preinvasive Ductal Carcinoma In Situ (DCIS) and very early breast cancer treated with anastrozole. To establish reduction in Ki-67 as a primary surrogate endpoint to breast cancer risk reduction in patients treated with anastrozole we will measure Ki-67 before and after treatment with anastrozole. Consistent with this, it has been demonstrated by Geisler et al that patients with advanced breast cancer show a decrease in Ki-67 on lumpectomy/mastectomy samples when anastrozole is administered for few weeks prior to definitive surgery. In addition, there is a trend for a more profound suppression in those achieving an objective response. Ki-67 will be measured by routine immunohistochemistry.

Specific Aim 2: We hypothesize that histopathological tumor response will be demonstrated in 30-40 percent of patients with preinvasive (DCIS) and early invasive (less than 2 cm) breast cancer treated with anastrozole. The percent ability to reverse early breast cancer lesions in patients treated with anastrozole will be qualified as a secondary surrogate endpoint to breast cancer risk reduction. Consistent with this, it has been demonstrated that 30-40 percent of patients with advanced breast cancer show an infiltration of foamy macrophages and fibrosis on lumpectomy/mastectomy samples when chemotherapy is administered for few months prior to definitive surgery. Further, there is a trend for a more profound change in those achieving a complete clinical response. Importantly, a complete pathological response in these advanced breast cancer has been shown to correlate with improved disease free survival and overall survival in breast cancer patients. A corollary is that if reversibility of early carcinogenic lesions is reliably demonstrated in our present proposal, it would translate into chemoprevention of breast cancer.

Specific Aim 3: To compare the pretreatment MRI with post treatment MRI (as a secondary surrogate endpoint to breast cancer risk reduction). We hypothesize that tumor response can be measured by contrast washout characteristic in patients with preinvasive and very early breast cancer treated with aromatase inhibitor. Consistent with this, we have previously demonstrated that patients with advanced breast cancer show a reduction in vascularity in response to chemotherapy. Further, there is a trend for a more profound suppression in those achieving a pathological response on lumpectomy/mastectomy specimen.

Specific Aim 4: To compare the pretreatment markers of angiogenesis with post treatment markers of angiogenesis (as a secondary surrogate endpoint to breast cancer risk reduction). We hypothesize that tumor response can be measured by reduction in CD31 (microvessel count), CD105 (endoglin) and VEGF in response to hormonal therapy. There may be upregulation of TSP-1, an angiogenesis inhibitor in response to anastrozole. Angiogenic activity has been reported for ligands of the nuclear hormone receptor superfamily such as estrogens. Inhibition of the proangiogenic effects of estrogens could underlie the chemopreventive action of hormone modulators on mammary carcinogenesis. A group of investigators have indeed coined the word angioprevention as a mechanism of chemoprevention that reverses the angiogenic switch from preinvasive to invasive cancer. Additionally, it has been demonstrated that patients with various cancers whose tumor vascularity is targeted with VEGF inhibitor show higher response than patients who are treated with chemotherapy alone. Our present proposal capitalizes on the data obtained in advanced breast cancer as to the efficacy of antiangiogenesis mechanism as an option in treatment and prevention .

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suspicion of DCIS or early invasive breast cancer on mammography.
* Patients must have histologically confirmed diagnosis of DCIS or early invasive breast cancer on core biopsy for final registration.
* Patients must be over 18 years of age
* "Patients must be postmenopausal as defined by one of the following criteria:

  1. Prior bilateral oophorectomy OR
  2. > 12 months since LMP with no prior hysterectomy OR
  3. a & b not applicable AND age >=50
* Patients must be positive for either ER or PR or both
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients must not have diagnosis of osteoporosis (T-score -2.5 according to the WHO)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-09-21 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mehta, MD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anastrozole
Started | 42
Completed | 34
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Anastrozole
Number analyzed (Participants) | 34
Age, Customized [Mean (Full Range); unit: years] | 63.2 [50 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Ki-67 Level
Time Frame: Baseline and up to 4 weeks
Population: 23 patients had both baseline data and off-treatment data available
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole
Number analyzed (Participants) | 23
Participants
  Decreased Ki-67 level | 15
  No Change in Ki-67 | 5
  Increased Ki-67 level | 3
Statistical Analysis 1: Comparison: Anastrozole; Test type: Other; p = 0.004, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 4.9, 95% CI 2-sided [1.8 to 8.0]

2. Secondary Outcome: Histopathological Response
Description: Assessed by changes in Nottingham grade
Time Frame: Baseline and up to 4 weeks
Population: 24 patients had baseline data and post-treatment available.
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole
Number analyzed (Participants) | 24
Participants
  Decreased | 7
  No Change | 17
Statistical Analysis 1: Comparison: Anastrozole; Test type: Other; p = 0.016, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.3, 95% CI 2-sided [0.10 to 0.49]

3. Secondary Outcome: To Compare Pretreatment Vascular Density With Post Treatment Vascular Density Using MRI
Time Frame: Baseline and 4 weeks after anastrozole
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole
Number analyzed (Participants) | 17
Participants
  Decreased | 7
  No Change | 9
  Increased | 1

4. Secondary Outcome: To Compare Pretreatment Markers of Angiogenesis With Post Treatment Marker of Angiogenesis
Time Frame: Baseline and up to 4 weeks
Population: Data was not collected and analysis of this outcome measure was not done.
Arm/Group | Anastrozole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First receipt of first of study drug until 30 days have elapsed following cessation of study drug, a total of up to 8 weeks.
Description: There were no reported serious adverse events for this trial.
Arm/Group | Anastrozole
All-Cause Mortality (participants affected / at risk) | 2/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 1/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=42)
Sores in mouth and between fingers (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2011-04-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT00256217/Prot_SAP_ICF_000.pdf